CLINICAL TRIAL: NCT01955954
Title: Investigation of the Canary Breathing System for Treating the Symptoms of Panic Disorder
Brief Title: Using the Canary Breathing System for Panic Disorder Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Health Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAHS 1-001-13
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Panic Disorder
Keywords: carbon dioxide monitoring; panic disorder; biofeedback; breathing training; Primary diagnosis; panic attacks
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Canary Breathing System (Experimental): Treatment with Canary Breathing System
  Interventions: Device: Canary Breathing System

INTERVENTIONS:
Device: Canary Breathing System — The Canary Breathing System is a biofeedback device meant to assist patients in the re-training of abnormal breathing patterns.

SUMMARY:
The purpose of this study is to test the effectiveness of the Canary Breathing System (CBS) in treating the symptoms of panic disorder.

DETAILED DESCRIPTION:
Panic disorder (PD) is associated with hyperventilation. The efficacy of a brief respiratory feedback program for PD has been previously established. The aim of the present study was to expand these results by testing a similar program with more clinically representative patients and settings. The intervention is delivered via home use following initial training by a clinician and provides remote monitoring of client adherence and progress by the clinician. Outcomes were assessed post-treatment and at 2- and 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Panic Disorder
* Subjects between 18 and 60 years of age (inclusive on day of enrollment)
* Subjects with a Clinician's Global Impression of > or = to 4.
* If on psychotropic medication, on a stable dose for a minimum of 3 months prior to enrollment
* If on psychotropic medication, an agreement to stay on their stable dose from study entry until the 2-month follow-up.

Exclusion Criteria:

* Pregnancy
* Current enrollment in another drug or device study
* Current enrollment in another drug or device study that is not at least 30 days past the final follow-up
* Currently undergoing cognitive behavioral therapy (or equivalent)
* Refractory to either a breathing training program or cognitive behavioral therapy (or equivalent) in the 3 months prior to enrollment
* Evidence of organic mental disorder
* Severe suicidality
* Presence of any psychotic disorder
* Bipolar disorder that is present for < 5 years; a major depressive, manic or hypomanic episode in the last 12 months; failure to take and maintain a stable dose of medication in treatment of bipolar disorder in the last 12 months
* Current alcohol or drug dependence
* Cardiovascular or pulmonary disease
* Epilepsy or seizures
* Undergoing additional psychologic treatment at any point from study enrollment to 2-month follow-up to treat panic disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Tolin, PhD, Principal Investigator — Institute of Living, Hartford Hospital
Locations (4):
- United States (4):
  - San Francisco Bay Area Center for Cognitive Therapy, Oakland, California
  - Institute of Living, Hartford, Connecticut
  - Alexian Brothers Center for Anxiety and OCD, Hoffman Estates, Illinois
  - Kansas City Center for Anxiety Treatment, P.A., Overland Park, Kansas

REFERENCES:
- [Result] Tolin DF, McGrath PB, Hale LR, Weiner DN, Gueorguieva R. A Multisite Benchmarking Trial of Capnometry Guided Respiratory Intervention for Panic Disorder in Naturalistic Treatment Settings. Appl Psychophysiol Biofeedback. 2017 Mar;42(1):51-58. doi: 10.1007/s10484-017-9354-4. PMID 28194546
- See also: Study Results — https://link.springer.com/content/pdf/10.1007%2Fs10484-017-9354-4.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Canary Breathing System
Started | 69
Received Treatment | 66
Completed Treatment | 53
Completed Post-treatment Assessement | 48
Completed 2-month Assessment | 46 (Primary endpoint)
Completed 6-month Assessement | 42
Completed | 33 (12-months)
Not Completed | 36

BASELINE CHARACTERISTICS:
Arm/Group | Canary Breathing System
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Achieving a 40% Decrease in Overall PDSS Score (Clinically Significant Response)
Description: The Panic Disorder Severity Scale (PDSS) (Shear, 1997) is a widely used assessment tool measuring panic disorder symptom severity and impact. Seven questions are scored from 0 to 4 giving minimum and maximum scores of zero and 28 respectively. Higher scores represent more severe impact of symptoms.
  A 40% decrease has been reported to be clinically significant (Furukawa et al 2009) and is defined as "Response" in this study.
Time Frame: Measured at 2 months post-treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Canary Breathing System
Number analyzed (Participants) | 46
Participants | 33

2. Secondary Outcome: Percent of Subjects Achieving a 40% Decrease in Overall PDSS Score (Clinically Significant Response)
Description: as for outcome 1
Time Frame: Measured post-treatment (week-5)
Measure: Count of Participants; unit: Participants
Arm/Group | Canary Breathing System
Number analyzed (Participants) | 48
Participants | 41

3. Secondary Outcome: Percent of Subjects Achieving a 40% Decrease in Overall PDSS Score (Clinically Significant Response)
Description: as for outcome 1
Time Frame: Measured at 12 months post-treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Canary Breathing System
Number analyzed (Participants) | 33
Participants | 27

4. Secondary Outcome: Percent of Subjects Achieving Zero Panic Attacks Reported in Previous Week
Time Frame: Measured post-treatment (week-5)
Measure: Count of Participants; unit: Participants
Arm/Group | Canary Breathing System
Number analyzed (Participants) | 48
Participants | 34

5. Secondary Outcome: Percent of Subjects Achieving Zero Panic Attacks Reported in Previous Week
Time Frame: Measured at 2 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Canary Breathing System
Number analyzed (Participants) | 46
Participants | 33

6. Secondary Outcome: Percent of Subjects Achieving Zero Panic Attacks Reported in Previous Week
Time Frame: Measured at 12 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Canary Breathing System
Number analyzed (Participants) | 33
Participants | 26

ADVERSE EVENTS:
Arm/Group | Canary Breathing System
All-Cause Mortality (participants affected / at risk) | 0/69
Serious Adverse Events (participants affected / at risk) | 0/69
Other Adverse Events (participants affected / at risk) | 1/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Canary Breathing System (N=69)
Dizziness (General disorders) | 1 (1)
Lightheadedness (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No